CLINICAL TRIAL: NCT03657316
Title: Impact of School Based Education Program on Dietary Knowledge, Attitude and Practice Among Preparatory School Girls in Assiut City
Brief Title: Impact of School Based Education Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dalia Atef, principle investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ISBEKAP
Record Dates: First submitted 2018-08-30; First posted 2018-09-05 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-08

CONDITIONS: Diet Modification
MeSH Terms: interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- experimental school 1 (Experimental): The experimental school 1 will receive the following:
  * Nutritional and physical activity educational workshop
  * Enhanced physical education
  * Involvement of the morning broadcast
  * Educational brochure will be sent to the parents
  * A monthly telephone call or a text message will be sent to the parents
  * Message to school administration to prevent selling of soft drinks and to sell healthy food
  * A monthly session (3 months)
  Interventions: Behavioral: nutrition education
- experimental school 2 (Experimental): The experimental school 2 school will receive a nutritional and physical activity educational workshop; that will be held on three days through one week; one hour session each day
  Interventions: Behavioral: nutrition education
- control (No Intervention): The control school will receive no intervention

INTERVENTIONS:
Behavioral: nutrition education — The content of the three days workshop:Healthy diet, Diet-related health risks and diseases, Physical activity The sustained multi-component program will be based on The three days nutritional and physical education workshop Enhanced physical education Involvement of the morning broadcast in provision of messages for students about nutrition and physical activity Brochure including key messages about diet and physical activity will be designed and sent to parents of the intervention classes of students A monthly telephone call or a text message will be sent to the parents to remind them about the commitment to the dietary health practices.
  Message to school administration to prevent selling of soft drinks and to sell healthy food A monthly session for three months will be held to remind the students with the messages
  Arms: experimental school 1; experimental school 2

SUMMARY:
Good health is an important indicator of the quality of life, in which healthy nutrition and physical activity take an important place. Healthy nutrition and physical activity according to the guidelines of WHO are closely related to lower general and speciﬁc mortality rates due to heart and coronary diseases and cancer, which are the top reasons for mortality from non-communicable diseases. Every year, 41 million people die from non-communicable diseases, which represents 71% of the total number of global deaths. This largely invisible epidemic is more serious in low- and middle-income countries, where 85% of non-communicable diseases premature deaths occur

DETAILED DESCRIPTION:
As unhealthy diet, physical inactivity and tobacco use are common risk factors of the non-communicable diseases, elimination of these modifiable risk factors would prevent 80% of premature heart disease, 80% of premature stroke, 80% of type 2 diabetes and 40% of cancer.

Studies indicate that good nutrition is especially important during adolescence, which is a period of biological and social change. These are crucial years for normal physical and mental development, and the diet and eating behaviors that develop during these years tend to persist throughout life. During adolescence, body size and composition, bodily functions and physical abilities change rapidly, and under-nutrition can slow height and weight growth and may delay puberty. In addition, healthful eating habits in young people not only help to prevent under-nutrition, growth retardation and acute nutritional problems, but also can enhance students' educational performance and learning . Nutrition-related health problems among the youth are apparent in developing countries where, paradoxically, both over- and under-nutrition can coexist.

At the global level, major modifications in the dietary habits have occurred since the second half of the twentieth century; first in industrial regions and more recently in developing countries. The concept of 'food' has changed from a means of nourishment to a marker of lifestyle and a source of pleasure as portrayed by media. A large proportion of televised food advertisements are of highly processed foods/convenient foods with, high caloric content, large amounts of fat and sugar, and with little or no micronutrient content .

Also, due to low cost and easy availability, people are increasingly consuming high-saturated-fat snacks, refined carbohydrates and sweetened carbonated beverages. There is an increased inclination to replace traditional meals with energy-dense imbalanced foods. Irregular meals, snacking, eating away from home, and following alternative dietary patterns have already been frequently reported among adolescents in many countries.

The traditional Egyptian diet has also been modified in the recent decades with introduction of new foods and eating habits.Such dietary patterns with inadequate physical activity trigger the onset of fat deposition and lead to early metabolic derangements such as the metabolic syndrome and type 2 diabetes mellitus .

A previous Egyptian study in Mansoura revealed unhealthy dietary habits of adolescents; as fast foods and carbonated drinks were consumed on daily bases by more than two thirds and one fifth of the participating students; respectively. It was also found that the majority of students drink tea more than 3 times daily. Excess salt and excess sugar/sweet intake were reported by more than half of the study participants.

Another study in the United Arab Emirates found that the majority of children and adolescent participants had less than the recommended number of servings from milk and vegetables.

A study in Saudi Arabia showed that large proportions of Saudi adolescent school students never consumed protein food sources or fresh fruits during the previous week, while the most frequently consumed food items were rice and bread.

Moreover, the majority of Arab adolescents do not meet the recommended guidelines for daily physical activity. It has been reported that more than 85% of girls and 75% of boys aged 13-15 years in seven Arab countries (Djibouti, Egypt, Jordan, Libya Morocco, Oman, and the United Arab Emirates) did not engage in a sufficient amount of daily physical activity (obtaining at least 60 minutes of physical activity per day).

A cross-cultural study on perceived barriers to healthy eating among adolescents in seven Arab countries revealed that there are several personal, social, and environmental barriers to healthy eating among adolescents in Arab countries; Lack of information on healthy eating, lack of motivation to eat healthy diets, and not having time to prepare or eat healthy foods due to school commitments were found to be the main barriers to healthy eating.

In order to promote healthier eating habits, nutrition knowledge is believed to be important. However, nutrition knowledge alone may not be sufficient to change dietary habits hence in addition there is need to mold a positive attitude toward healthy eating early in childhood. With the current change in dietary habits to the western diet and increase in televised food advertisements targeting children, there is even greater need to empower children with the right knowledge and attitudes for making proper food choices. There is a growing evidence suggesting that young children from developing countries are increasingly making unhealthy food choices especially due to lack of knowledge and wrong perception towards healthy foods.

However, children do not always choose what they eat; very often parents decide and prepare food for them. Clearly, parents, peers and teachers can play a crucial role in shaping each child's outlook towards health.

Nutrition knowledge alone does not influence behavior, but does provide individuals with the ability to know how to select a healthy diet. The nutritional knowledge and skills need to be taught during childhood when firm eating practices are being established. Therefore, school is the major area for providing young people with nutrition knowledge and skills.

Some previous studies revealed that school based nutritional education programs resulted in significant positive changes in both nutrition knowledge and behaviors, while other studies revealed non-significant changes.

Strategies are more effective when they include efforts to increase parental or family support. Family involvement enhances the effectiveness of programs for younger children. Objectives for the family component in successful programs focus on stimulating awareness and gaining parental support to encourage variety in the diet and availability of healthy foods at home. Methods used include brochures and activities with the Parents' Association and the Parent-Teachers' Association.

Environmental interventions are important components of intervention programs, that contribute to the creation of opportunities for action by removing barriers to following a healthy diet.

School-based nutrition education should address the needs and interests of students, the teachers and the school; take into account what children already know and can do; be culturally appropriate; be delivered in a way children can understand and teach the skills and knowledge required to improve or strengthen healthy eating habits. Several studies have shown that using different teaching and learning strategies can enhance the learning outcomes of school children as small group discussions, group work, demonstrations, art educational drawing help in the success of the intervention program.

Efficacy of nutrition education interventions also depends on the duration and frequency of intervention. Two systematic review concluded that educational interventions that are sustained for a longer are more likely to be effective than those conducted for a short period. Adequate time, intensity of the intervention, resources, as well as the provision of suitable materials and teacher training opportunities are essential to program success. Moreover having support from policy makers and school management affect the success of the program.

ELIGIBILITY:
Inclusion Criteria:

* Second year preparatory school female students in Assiut city.
* A group of female preparatory school students' mothers will be invited to participate in focus groups discussions from each school.

Exclusion Criteria:

-

Ages: 11 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 270 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Dietary knowledge | 5 months after the start of the intervention. immediately after end of the sustainable program
  The level of nutrition knowledge will be determined using questions concerning nutrients and their functions, food sources, dietary needs and concept of balanced diet, healthy eating, diet-related health risks and diseases. Knowledge score will be calculated The level of nutrition knowledge will be determined using questions concerning nutrients and their functions, food sources, dietary needs and concept of balanced diet, healthy eating, diet-related health risks and diseases.
  • Nutrition attitude: Nutrition attitude will be assessed through questions including attitudes towards the importance of nutrition and developing healthy dietary habits. The subjects will be asked to state their level of agreement or disagreement with statements using a Likert scale.
  • Dietary practices: Dietary practices will be evaluated through food frequency questionnaire and questions on some dietary habits as regularity of meals and main type of snacks.
Nutrition attitude | 5 months after the start of the intervention. immediately after end of the sustainable program
  Nutrition attitude will be assessed through questions including attitudes towards the importance of nutrition and developing healthy dietary habits. The subjects will be asked to state their level of agreement or disagreement with statements using a Likert scale. Attitude score will be calculated
Dietary practices | 5 months after the start of the intervention. immediately after end of the sustainable program
  Dietary practices will be evaluated through food frequency questionnaire and questions on some dietary habits as regularity of meals and main type of snacks

SECONDARY OUTCOMES:
Body mass index | 5 months after the start of the intervention. immediately after end of the sustainable program
  Weight will be measured by the nearest 0.1 kg using a portable digital scale. A portable stadiometer will be used to obtain height measurements to the nearest 0.1 cm. Body mass index (BMI) will be calculated using the standard formula (kg/m2). BMI percentile will be used to classify weight status (i.e., underweight, normal weight, overweight, and obese)

CONTACTS AND LOCATIONS:
Overall Officials: Dalia Mohamed Atef Shehata, MSC, Principal Investigator — Assiut University
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Collins CE, Dewar DL, Schumacher TL, Finn T, Morgan PJ, Lubans DR. 12 month changes in dietary intake of adolescent girls attending schools in low-income communities following the NEAT Girls cluster randomized controlled trial. Appetite. 2014 Feb;73:147-55. doi: 10.1016/j.appet.2013.11.003. Epub 2013 Nov 12. PMID 24239513
- [Background] Ali HI, Ng SW, Zaghloul S, Harrison GG, Qazaq HS, El Sadig M, Yeatts K. High proportion of 6 to 18-year-old children and adolescents in the United Arab Emirates are not meeting dietary recommendations. Nutr Res. 2013 Jun;33(6):447-56. doi: 10.1016/j.nutres.2013.03.008. Epub 2013 May 4. PMID 23746560
- [Background] Amaya-Castellanos C, Shamah-Levy T, Escalante-Izeta E, Morales-Ruan Mdel C, Jimenez-Aguilar A, Salazar-Coronel A, Uribe-Carvajal R, Amaya-Castellanos A. Development of an educational intervention to promote healthy eating and physical activity in Mexican school-age children. Eval Program Plann. 2015 Oct;52:159-68. doi: 10.1016/j.evalprogplan.2015.05.002. Epub 2015 Jun 11. PMID 26099561
- [Background] Fahlman MM, Dake JA, McCaughtry N, Martin J. A pilot study to examine the effects of a nutrition intervention on nutrition knowledge, behaviors, and efficacy expectations in middle school children. J Sch Health. 2008 Apr;78(4):216-22. doi: 10.1111/j.1746-1561.2008.00289.x. PMID 18336681
- [Background] Hassan-Wassef H. Food habits of the Egyptians: newly emerging trends. East Mediterr Health J. 2004 Nov;10(6):898-915. PMID 16335778
- [Background] Murimi MW, Kanyi M, Mupfudze T, Amin MR, Mbogori T, Aldubayan K. Factors Influencing Efficacy of Nutrition Education Interventions: A Systematic Review. J Nutr Educ Behav. 2017 Feb;49(2):142-165.e1. doi: 10.1016/j.jneb.2016.09.003. Epub 2016 Nov 1. PMID 27814976
- [Background] Musaiger AO, Al-Mannai M, Tayyem R, Al-Lalla O, Ali EY, Kalam F, Benhamed MM, Saghir S, Halahleh I, Djoudi Z, Chirane M. Perceived barriers to healthy eating and physical activity among adolescents in seven Arab countries: a cross-cultural study. ScientificWorldJournal. 2013 Nov 14;2013:232164. doi: 10.1155/2013/232164. eCollection 2013. PMID 24348144
- [Background] Perez-Rodrigo C, Aranceta J. School-based nutrition education: lessons learned and new perspectives. Public Health Nutr. 2001 Feb;4(1A):131-9. doi: 10.1079/phn2000108. PMID 11255503
- [Background] Shah P, Misra A, Gupta N, Hazra DK, Gupta R, Seth P, Agarwal A, Gupta AK, Jain A, Kulshreshta A, Hazra N, Khanna P, Gangwar PK, Bansal S, Tallikoti P, Mohan I, Bhargava R, Sharma R, Gulati S, Bharadwaj S, Pandey RM, Goel K. Improvement in nutrition-related knowledge and behaviour of urban Asian Indian school children: findings from the 'Medical education for children/Adolescents for Realistic prevention of obesity and diabetes and for healthy aGeing' ( MARG) intervention study. Br J Nutr. 2010 Aug;104(3):427-36. doi: 10.1017/S0007114510000681. Epub 2010 Apr 7. PMID 20370939